CLINICAL TRIAL: NCT02291692
Title: Ultrasound Guided Thoracic Paravertebral Block
Brief Title: Ultrasound Guided Thoracic Paravertebral Block for Percutaneous Nephrolithotomy Operations in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Zehra, Zehra Hatipoglu, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PVB
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paravertebral blockade (Active Comparator): Paravertebral blockade
  Interventions: Procedure: paravertebral blockade
- Paracetamol (No Intervention): The patients was given 15 mg/kg of paracetamol.

INTERVENTIONS:
Procedure: paravertebral blockade — ultrasound guided thoracic paravertebral block with 0.5 ml/kg bupivacaine %0.5
  Arms: Paravertebral blockade

SUMMARY:
The investigators aimed to evaluate the effect of ultrasound guided thoracic paravertebral block with bupivacaine on both perioperative anesthetic agent consumption and postoperative analgesia in pediatric patients undergoing percutaneous nephrolithotomy for kidney stone.

DETAILED DESCRIPTION:
This study was performed after approval of Ethics Committee and parents written consent. Between the ages 1-5, planned percutaneous nephrolithotomy due to kidney stones 40 patients were enrolled in this study, and patients were randomly divided into two group. All patients were performed general anaesthesia. The Group I patients was given ultrasound guided thoracic paravertebral block with 0.5 ml/kg bupivacaine %0.5 after giving prone position and the Group II patients was given 15 mg/kg of paracetamol as postoperative analgesia. In the period of postoperative, if the FLACC > 4; it was planned to dose 1 mg/kg of tramadol. Patients' hemodynamic parameters, oxygen saturation, sevoflurane concentration were recorded 10, 15, 30 and 60 minutes intraoperatively. Patients' hemodynamic parameters, oxygen saturation, pain scores (FLACC), satisfaction of parents, the number of patients who additional analgesic requirements and side effects (nausea,vomiting, hypotension, bradycardia, respiration problems etc) were recorded in the postoperative period. Primary outcome measures was pain scores using FLACC scale.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* Between the ages of 1-5 years
* Forty children

Exclusion Criteria:

* Refusals by parents
* Children with spine deformities
* Cutaneous infection
* Bleeding diathesis
* Allergy to drugs used
* ASA physical status III-IV

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain score | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Akıncı, MD, Principal Investigator — Cukurova University

REFERENCES:
- [Background] Berta E, Spanhel J, Smakal O, Smolka V, Gabrhelik T, Lonnqvist PA. Single injection paravertebral block for renal surgery in children. Paediatr Anaesth. 2008 Jul;18(7):593-7. doi: 10.1111/j.1460-9592.2008.02592.x. Epub 2008 May 8. PMID 18482238